CLINICAL TRIAL: NCT02392988
Title: Randomised ,Single Blind, Placebo Controlled in Meir Medical Center. Study the Potential of Acupuncture Therapy to Reduce the Need for Labor Induction After Postdate (Week 41)
Brief Title: Does Acupuncture Therapy Reduce the Need for Labor Induction After Postdate (Week 41)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Clalit Health Services (Other); Reidman college (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0002-15
Record Dates: First submitted 2015-03-02; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-02

CONDITIONS: Post-term Pregnancy (40 to 42 Weeks Gestation)
MeSH Terms: conditions — Pregnancy, Prolonged | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group receives sham treatment (Placebo Comparator): Sham treatment will be given on points on the back, points that are not acupuncture points, so that the patient will not be able to know whether she is receiving sham treatment or a real treatment. The treatment will be every 48-72 hours, a maximum of three treatments.
  Interventions: Other: Placebo Comparator
- Group receives acupuncture treatment (Experimental): The women in this group will receive acupuncture treatment every 48-72 hours, a maximum of three treatments.
  Interventions: Other: acupuncture treatment
- Group doesn't receive any treatment (No Intervention): The women in this group will come for a follow-up check a week later, unless a spontaneous birth will develop.

INTERVENTIONS:
Other: acupuncture treatment — acupuncture treatment
  Arms: Group receives acupuncture treatment
Other: Placebo Comparator — Placebo Comparator
  Arms: Group receives sham treatment

SUMMARY:
In recent years, it is accepted to induce birth at week 41 in order to reduce the risk in surplus pregnancies. It was found that after 41 weeks, there is a significant increase in pregnancy complications including meconium liquor, shoulder dystocia and fetal death in uterus.

Induction at 41 weeks was found to reduce the risk of complications described above, without taking the risk of cesarean section and, therefore, the recommendation of the Israel Society of Maternal Fetal Medicine, is to induce birth for women who completed 41 weeks of pregnancy.

Induction is performed mechanically by entering a balloon to the cervix or by medicated prostaglandins and later, intravenous Pitocin to most women. The process takes two to three days with about 60-70% success rate.

In recent years there has been a growing awareness to use natural methods to start labor.

Many women tend to turn to natural medicine in order to reduce the need for conventional drugs to start labor.

Given the lack of research on the issue and considering the rising demand of the involvement of alternative medicine in labor induction process, the investigators decided to carry out research on this subject.

DETAILED DESCRIPTION:
To the study will be recruited women who have completed 40 weeks of pregnancy and have not yet given birth, with proper evaluation of mother and fetus.

Women who are fit to participate and had given their consent, will be computerized randomized to one of three groups.

Research groups:

1. Group who receives acupuncture treatment in order to accelerate the development of birth.
2. Group who receives sham treatment - non acupuncture treatment, but a similar treatment, so that the patient is unable to know whether she is receiving a real acupuncture treatment, or the similar one, which has no effect on the patient.
3. Group who does not receive any treatment and will be reviewed a week later, unless a spontaneous birth will be developed. (Procedure accepted today) The study will be carried out between week 40 and week 41. During the week acupuncture treatment, sham treatment or conservative follow-up will be carried out, depending on the study group differentiation.

All women who will be randomized to the treatment groups, will fill a preliminary questionnaire for acupuncture treatment.

The course of treatment: During the week of study the women in the treatments groups will receive treatment every 48-72 hours, a maximum of three treatments.

Measures will be taken on the following week or two when the women will come to give birth.

ELIGIBILITY:
Inclusion Criteria:

1. Women past their due date (week 40)
2. Proper dating of pregnancy
3. Uncomplicated pregnancy
4. Normal evaluation as part of the mother and fetus routine examination on week 40
5. Singleton pregnancy
6. No contraindication for vaginal birth
7. No significant signs of birth

Exclusion Criteria:

1. Past Cesarean Section
2. Women who have undergone acupuncture treatment during pregnancy
3. Women who did not undergo separation membranes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The number of women who received birth induction after week 41 | three weeks

SECONDARY OUTCOMES:
Number of women who had SROM (spontaneous rupture of membranes) or AROM (artificial rupture of membranes). | three weeks
Duration of labour | three weeks
Time past from treatment (acupuncture vs. placebo) till labour | three weeks
Hg before and after labour | three weeks
Number of women who received epidural | three weeks
Type of labour | three weeks
Apgar score after birth | three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tal Biron-Shental, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medial Center, Kfar Saba, Israel